CLINICAL TRIAL: NCT01767363
Title: Prostate Cancer in Benign Prostatic Hyperplasia (BPH) Patients
Brief Title: WEUSKOP5723: Prostate Cancer Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116059; WEUSKOP5723 (Other: GSK)
Record Dates: First submitted 2012-12-19; First posted 2013-01-14 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Prostatic Hyperplasia
Keywords: 5-alpha reductase inhibitor; benign prostatic hyperplasia treatment; Prostate cancer mortality
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — 5-alpha Reductase Inhibitors; Adrenergic alpha-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 5-alpha reductase inhibitors with or without alpha-blockers: Men using 5-alpha reductase inhibitors with or without alpha-blockers over the course of the study period.
  Interventions: Other: 5-alpha reductase inhibitors; Other: Alpha-blockers
- Alpha-blockers: Men using alpha-blockers over the course of the study period.
  Interventions: Other: 5-alpha reductase inhibitors; Other: Alpha-blockers

INTERVENTIONS:
Other: 5-alpha reductase inhibitors — Use of 5-alpha reductase inhibitors over the course of the study period.
Other: Alpha-blockers — Use of alpha-blockers over the study period.

SUMMARY:
This retrospective cohort study will assess the association of benign prostatic hyperplasia (BPH) treatment (5-alpha reductase inhibitors (5ARI) and alpha-blocker medications) with the occurrence of prostate cancer related mortality. This study will also assess a number of secondary endpoints including prostate cancer mortality or metastatic prostate cancer, and all cause mortality.

DETAILED DESCRIPTION:
A retrospective cohort study from 1992-2010 will be conducted using data from 4 Kaiser sites: Kaiser Permanente Southern California (KPSC), Kaiser Permanente Northern California (KPNC), Kaiser Permanente Northwest (KPNW), and Kaiser Permanente Colorado (KPCO). Men treated with BPH medications, 5ARIs (with and without concomitant and/or previous alpha-blocker use) will be compared to men treated with alpha-blockers. A matched design will be used with each man treated with 5ARIs being matched with 5 or 6 men treated with alpha-blockers. Men 50 years or older at the time of their first prescription for a study defined BPH medication, initiating treatment between 1992 and 2008 with at least 1-year of coverage in the healthcare system before the first prescription for BPH medication and at least 3 consecutive prescriptions (90 days of supply) for a BPH medication will be eligible for inclusion in the study. Men with a diagnosis of prostate cancer any time before the first prescription for BPH medication, having a diagnosis of prostate cancer within 3 months after initiation of their first BPH medication, and those treated with finasteride 1mg prior to their BPH medication will be excluded from the study. 5ARI initiators will be matched to alpha-blocker users in a ratio of 1:5 or 1:6 to yield an overall matching ratio of 1:5.4. Matching factors include age (+/- 1 year), timing of BPH treatment initiation (+/- 1 year), race, and duration of prior use of alpha-blockers. Based on the feasibility study from KPSC, there will be approximately 284,000 men treated with BPH medications meeting eligibility criteria for inclusion in the study sample.

The data will be analyzed using Kaplan Meier curves comparing the 5ARI vs alpha-blocker users for the primary and secondary study outcomes, without any adjustments. Additionally, a plot of cumulative incidence, adjusting for competing risks of death, will be constructed allowing for the investigation of the effect of competing risks on the Kaplan-Meier probability estimates. Crude mortality rates and incidence rates of metastatic cancer will be calculated. Cox proportional hazard regression models will be fit to compare the primary and secondary outcomes between groups using hazard ratios, while adjusting for pre-treatment characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are Male
* Patients that have a new prescription for BPH medication (5ARI and/or alpha-blocker) in 1992 or later that is identified as appropriate treatment for BPH/LUTS from the KP National Pharmacy guidelines.
* Patients with a treatment with BPH medication must be initiated prior to Jan1, 2008.
* Patients age 50 years or older at time of treatment with 5ARI or alpha-blocker.
* Patients with at least 1-year of coverage in the healthcare system before the first prescription for BPH medication (5ARI and/or alpha-blocker).
* Patients with at least 3 consecutive prescriptions (90 days of supply) for a BPH medication (5ARI and/or alpha-blocker).

Exclusion Criteria:

* Patients with a diagnosis of prostate cancer any time before the first prescription for BPH medication (5ARI and/or alpha-blocker).
* Patients with a dagnosis of prostate cancer within 3 months after first BPH medication (5ARI and/or alpha-blocker)
* Patients treated with Finasteride 1mg prior to BPH medication. Finasteride 1mg is the dose approved for androgenic alopecia and as the target population for this study is men with treated BPH, we will exclude all men treated with the 1mg dose.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All men age 50 years and older treated with a BPH medication (5ARI and/or alpha-blocker) will be eligible for inclusion. Participants are not required to have a BPH diagnosis at the time of their first 5ARI or alpha-blocker prescription as based upon data from the feasibility report approximately half of all men received their first recorded BPH diagnosis after initiating treatment. Furthermore, approximately 25% of participants treated with 5ARIs or alpha-blockers did not have a diagnosis code for BPH in their medical record. BPH diagnosis codes were not used in a consistent way historically in the Kaiser data. Men should have coverage within the healthcare system for at least 1-year before the first BPH medication prescription. Men with a history of prostate cancer or who develop prostate cancer within <3 months of starting their first BPH medication are not eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is prostate cancer related mortality. | 17 years
  Cause of death codes from death certificates, along with an electronic algorithm using pre-defined decision points, will be used to classify cause of death. Chart review will be performed to further validate cause of death.

SECONDARY OUTCOMES:
One of the secondary outcomes is all cause mortality. Death information will be derived from several sources including membership files, state death records and the Social Security Index. | 17 years
One of the secondary outcomes is the combined endpoint of prostate cancer mortality or metastatic prostate cancer. | 17 years
  Metastatic prostate cancer will be identified using data recorded in cancer registries and with an algorithm based on patient medical records.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline